CLINICAL TRIAL: NCT01825135
Title: Electrical Stimulation to Strengthen the Quadriceps Muscles in Patients Requiring Prolonged Mechanical Ventilation
Brief Title: Electrical Stimulation to Strengthen Muscles in the Lower Legs in Patients Requiring Prolonged Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RML Specialty Hospital (Other)
Responsible Party: Principal Investigator, Amal Jubran, Principle Investigator-Staff Physician, RML Specialty Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXJ012
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Muscle Weakness
Keywords: muscle strength; muscle function; functional status
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular electrical stimulation (Experimental): Neuromuscular electrical stimulation (NMES) will be applied to the quadriceps muscles for 30 minutes
  Interventions: Device: Neuromuscular electrical stimulation
- Sham stimulation (Sham Comparator): Sham stimulation will be applied to the quadriceps for 30 minutes
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation
  Other Names: 300PV™ neuromuscular stimulation (NMES)device
  Arms: Neuromuscular electrical stimulation
Device: sham stimulation — sham stimulation will be applied to the quadriceps
  Other Names: 300PV™ Neuromuscular Stimulation (NMES) device
  Arms: Sham stimulation

SUMMARY:
The primary aim of this proposal is to test the effectiveness of NMES in improving functional status and muscle function in patients requirng prolonged mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* duration of mechanical ventilation for 14 days or more
* sufficiently awake
* able to speak and comprehend English

Exclusion Criteria:

* known primary neuromuscular disease
* lower extremities paresis or amputee
* patients with left-ventricular assist device (LVAD)
* cardiopulmonary instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
modified Functional Independence Measurement (FIM) score | Hospital discharge, an expected average stay of 5 weeks
  Functional status as measured by modified Functional Independence Measurement (FIM) score

CONTACTS AND LOCATIONS:
Overall Officials: Amal Jubran, MD, Principal Investigator — RML Specialty Hospital
Locations (1):
- RML Specialty Hospital, Hinsdale, Illinois, United States